CLINICAL TRIAL: NCT05500183
Title: Evaluating the Effects of a Cognitively Enriched Walking Program for Older Adults on Cognitive Functioning, Psychosocial Wellbeing and Physical Activity: a Randomized Controlled Trial
Brief Title: Cognitively Enriched Walking Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WALKYOURBRAIN
Record Dates: First submitted 2022-07-08; First posted 2022-08-15 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy Aging; Cognitive Decline; Physical Inactivity
MeSH Terms: conditions — Cognitive Dysfunction; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PA + CA (Experimental): a cognitively enriched walking program (Physical Activity (PA)+Cognitive Activity (CA)
  Interventions: Behavioral: Cognitively enriched walking program
- PA only (Active Comparator): a walking program without cognitive enrichment (Physical Activity (PA) only)
  Interventions: Behavioral: walking program
- control (No Intervention): a passive control group (CG). The passive CG will receive no intervention program.

INTERVENTIONS:
Behavioral: Cognitively enriched walking program — The PA+CA program is group-based and will have a duration of six months (i.e. 24 weeks), with a frequency of two group sessions a week. All group sessions will last for approximately one hour and take place in groups of twelve or thirteen people supervised by a certified coach. Participants will be encouraged to do one individual session every week, as well.
  Arms: PA + CA
Behavioral: walking program — The PA only program is group-based and will have a duration of six months (i.e. 24 weeks), with a frequency of two group sessions a week. All group sessions will last for approximately one hour and take place in groups of twelve or thirteen people supervised by a certified coach. Participants will be encouraged to do one individual session every week, as well.
  Arms: PA only

SUMMARY:
Dementia currently affects more than 47 million people worldwide, its prevalence is forecasted to triple by 2050, and it has been reported to be one of the most costly disorders in Belgium. There is good scientific evidence that the cognitive impairments associated with the development of dementia can be lessened or even reversed thanks to the plasticity of the brain (rewiring). Recent research has shown that physical activity combined with performing cognitively challenging tasks is a very potent way to induce this rewiring of the brain, which can enable people to improve their cognitive functions. Yet, so far, these studies are mainly limited to controlled laboratory conditions. The investigators developed a real-life cognitively enriched walking program, with input from experts and end-users. In this study, the investigators will examine the added value of enriching physical activity (walking) with cognitive exercises in improving cognition of older adults by conducting a six-month community-based randomized controlled trial. The investigators will also examine the longer term effectiveness in a follow-up measurement visit six months after the program. The investigators will focus on the following outcomes: cognitive functioning (i.e., objective, subjective and cognitive activity), psychosocial wellbeing (i.e., loneliness, social support, depressive symptomatology, positive wellbeing and expectations regarding aging), physical activity (i.e. both objective and subjective) and general health.

ELIGIBILITY:
Inclusion Criteria:

1. male and female volunteers
2. aged 65 years and older
3. community-dwelling

Exclusion Criteria:

1. Have a neurodegenerative disorder (i.e. Alzheimer's disease, Parkinson's disease, Multiple Sclerosis,…);
2. Are diagnosed with mild cognitive impairment (MCI);
3. Are diagnosed with a psychiatric disorder (e.g. schizophrenia, bipolar disorder, borderline personality disorder,…);
4. Are currently having a depressive episode;
5. Have had a serious brain injury in the past year, or before and still experience consequences (i.e. traumatic brain injury, stroke, brain haemorrhage);
6. Have a history of, or current, addiction to drugs or excessive alcohol abuse;
7. Are not able to walk approximately three kilometres in one hour (at an average walking pace);
8. Make use of a walking aid (i.e. a cane, a (rollator) walker, or a wheelchair);
9. One or both of their parents were diagnosed with juvenile dementia;
10. Know in advance that they will not be will not be present for one or more periods of longer than one month (e.g. because of a long holiday).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
objective cognitive functioning T1 | baseline
  - Cambridge Neuropsychological Test Automated Battery (CANTAB) (Bento-Torres et al., 2017; Sahakian & Owen, 1992; Zygouris & Tsolaki, 2015): objective cognitive functioning is assessed with CANTAB. Different tests can be configured in a test battery, based on the focus of the study. The tests are non-verbal and culturally independent and make use of touchscreen technology. The CANTAB has been shown sensitive to changes in cognitive performance. Six different tests were selected to obtain a comprehensive view of one's objective cognitive functioning. The selected tests assess attention (i.e. sustained attention), memory (i.e. visual episodic attention and short term visual memory) and executive functioning (i.e. working memory and strategy).
objective cognitive functioning T2 | 3 months follow-up
  - Cambridge Neuropsychological Test Automated Battery (CANTAB) (Bento-Torres et al., 2017; Sahakian & Owen, 1992; Zygouris & Tsolaki, 2015): objective cognitive functioning is assessed with CANTAB. Different tests can be configured in a test battery, based on the focus of the study. The tests are non-verbal and culturally independent and make use of touchscreen technology. The CANTAB has been shown sensitive to changes in cognitive performance. Six different tests were selected to obtain a comprehensive view of one's objective cognitive functioning. The selected tests assess attention (i.e. sustained attention), memory (i.e. visual episodic attention and short term visual memory) and executive functioning (i.e. working memory and strategy).
objective cognitive functioning T3 | 6 months follow-up
  - Cambridge Neuropsychological Test Automated Battery (CANTAB) (Bento-Torres et al., 2017; Sahakian & Owen, 1992; Zygouris & Tsolaki, 2015): objective cognitive functioning is assessed with CANTAB. Different tests can be configured in a test battery, based on the focus of the study. The tests are non-verbal and culturally independent and make use of touchscreen technology. The CANTAB has been shown sensitive to changes in cognitive performance. Six different tests were selected to obtain a comprehensive view of one's objective cognitive functioning. The selected tests assess attention (i.e. sustained attention), memory (i.e. visual episodic attention and short term visual memory) and executive functioning (i.e. working memory and strategy).
cognitive functioning T4 | 12 months follow-up
  - Cambridge Neuropsychological Test Automated Battery (CANTAB) (Bento-Torres et al., 2017; Sahakian & Owen, 1992; Zygouris & Tsolaki, 2015): objective cognitive functioning is assessed with CANTAB. Different tests can be configured in a test battery, based on the focus of the study. The tests are non-verbal and culturally independent and make use of touchscreen technology. The CANTAB has been shown sensitive to changes in cognitive performance. Six different tests were selected to obtain a comprehensive view of one's objective cognitive functioning. The selected tests assess attention (i.e. sustained attention), memory (i.e. visual episodic attention and short term visual memory) and executive functioning (i.e. working memory and strategy).
subjective cognitive functioning T1 - Cognitive Failures Questionnaire | baseline
  Cognitive Failures Questionnaire (CFQ) (Broadbent et al., 1982; Ponds et al., 2006): this self-administered questionnaire assesses subjective cognitive functioning. Participants are asked about minor everyday slips or errors. It is not a replacement for testing objective cognitive functioning, but reflects the experience of the frequency of everyday slips of the participant.
  The CFQ consists of 25 items. Participants have to rate the items on a five-point response scale going from "1" (very ofen) to "5" (never). Higher scores reflect less cognitive failure.
subjective cognitive functioning T1 - Cognitive and Leisure Activities Scale (CLAS) | baseline
  Cognitive and Leisure Activities Scale (CLAS) (Galvin et al., 2021): this is a measure of the type and frequency of cognitive activities. It includes sixteen types of cognitive activities and is self-administered. Even though it is difficult to establish the validity of this new questionnaire since there is no gold standard to measure cognitive activity, it is suggested that this questionnaire has a good content validity.
  The CLAS consists of 16 items that are scored on a five-point response scale, going from 0 "never" to 5 "daily". Higher scores reflect a higher frequency of doing the activity.
subjective cognitive functioning T2 - Cognitive Failures Questionnaire (CFQ) | 3 months follow-up
  Cognitive Failures Questionnaire (CFQ) (Broadbent et al., 1982; Ponds et al., 2006): this self-administered questionnaire assesses subjective cognitive functioning. Participants are asked about minor everyday slips or errors. It is not a replacement for testing objective cognitive functioning, but reflects the experience of the frequency of everyday slips of the participant.
subjective cognitive functioning T2 - Cognitive and Leisure Activities Scale (CLAS) | 3 months follow-up
  Cognitive and Leisure Activities Scale (CLAS) (Galvin et al., 2021): this is a measure of the type and frequency of cognitive activities. It includes sixteen types of cognitive activities and is self-administered. Even though it is difficult to establish the validity of this new questionnaire since there is no gold standard to measure cognitive activity, it is suggested that this questionnaire has a good content validity.
  The CLAS consists of 16 items that are scored on a five-point response scale, going from 0 "never" to 5 "daily". Higher scores reflect a higher frequency of doing the activity.
subjective cognitive functioning T3 - Cognitive Failures Questionnaire (CFQ) | 6 months follow-up
  Cognitive Failures Questionnaire (CFQ) (Broadbent et al., 1982; Ponds et al., 2006): this self-administered questionnaire assesses subjective cognitive functioning. Participants are asked about minor everyday slips or errors. It is not a replacement for testing objective cognitive functioning, but reflects the experience of the frequency of everyday slips of the participant.
  The CFQ consists of 25 items. Participants have to rate the items on a five-point response scale going from "1" (very ofen) to "5" (never). Higher scores reflect less cognitive failure.
subjective cognitive functioning T3 - Cognitive and Leisure Activities Scale (CLAS) | 6 months follow-up
  Cognitive and Leisure Activities Scale (CLAS)(Galvin et al., 2021): this is a measure of the type and frequency of cognitive activities. It includes sixteen types of cognitive activities and is self-administered. Even though it is difficult to establish the validity of this new questionnaire since there is no gold standard to measure cognitive activity, it is suggested that this questionnaire has a good content validity.
  The CLAS consists of 16 items that are scored on a five-point response scale, going from 0 "never" to 5 "daily". Higher scores reflect a higher frequency of doing the activity.
subjective cognitive functioning T4 - Cognitive Failures Questionnaire (CFQ) | 12 months follow-up
  Cognitive Failures Questionnaire (CFQ) (Broadbent et al., 1982; Ponds et al., 2006): this self-administered questionnaire assesses subjective cognitive functioning. Participants are asked about minor everyday slips or errors. It is not a replacement for testing objective cognitive functioning, but reflects the experience of the frequency of everyday slips of the participant.
  The CFQ consists of 25 items. Participants have to rate the items on a five-point response scale going from "1" (very ofen) to "5" (never). Higher scores reflect less cognitive failure.
subjective cognitive functioning T4 - Cognitive and Leisure Activities Scale (CLAS) | 12 months follow-up
  Cognitive and Leisure Activities Scale (CLAS) (Galvin et al., 2021): this is a measure of the type and frequency of cognitive activities. It includes sixteen types of cognitive activities and is self-administered. Even though it is difficult to establish the validity of this new questionnaire since there is no gold standard to measure cognitive activity, it is suggested that this questionnaire has a good content validity.
  The CLAS consists of 16 items that are scored on a five-point response scale, going from 0 "never" to 5 "daily". Higher scores reflect a higher frequency of doing the activity.

SECONDARY OUTCOMES:
Psychosocial wellbeing questionnaires T1 | baseline
  (i.e., loneliness, social support, depressive symptomatology, positive wellbeing and expectations regarding aging)
Psychosocial wellbeing questionnaires T2 | 3 months follow-up
  (i.e., loneliness, social support, depressive symptomatology, positive wellbeing and expectations regarding aging)
Psychosocial wellbeing questionnaires T3 | 6 months follow-up
  (i.e., loneliness, social support, depressive symptomatology, positive wellbeing and expectations regarding aging)
Psychosocial wellbeing questionnaires T4 | 12 months follow-up
  (i.e., loneliness, social support, depressive symptomatology, positive wellbeing and expectations regarding aging)
Physical activity assessment (subjective) T1 | baseline
  International Physical Activity Questionnaire - Short Form (IPAQ-SF) (Craig et al., 2003): this is an extensively used self-report measure for physical activity during the past seven days. It provides us with a categorical score of physical activity, distinguishing between low, moderate and high levels of physical activity.
Physical activity assessment (objective) T1 | baseline
  Actigraph accelerometer at hip (Barnett et al., 2016): this is an objective measure of physical activity level, frequently used in physical activity studies with older adults. Participants will be asked to wear this accelerometer during seven days (day and night). They will be asked to register when and why they did not wear the device in a personal diary provided by the researchers.
Physical activity assessment (subjective) T2 | 3 months follow-up
  International Physical Activity Questionnaire - Short Form (IPAQ-SF) (Craig et al., 2003): this is an extensively used self-report measure for physical activity during the past seven days. It provides us with a categorical score of physical activity, distinguishing between low, moderate and high levels of physical activity.
Physical activity assessment (objective) T2 | 3 months follow-up
  Actigraph accelerometer at hip (Barnett et al., 2016): this is an objective measure of physical activity level, frequently used in physical activity studies with older adults. Participants will be asked to wear this accelerometer during seven days (day and night). They will be asked to register when and why they did not wear the device in a personal diary provided by the researchers.
Physical activity assessment (subjective) T3 | 6 months follow-up
  International Physical Activity Questionnaire - Short Form (IPAQ-SF) (Craig et al., 2003): this is an extensively used self-report measure for physical activity during the past seven days. It provides us with a categorical score of physical activity, distinguishing between low, moderate and high levels of physical activity.
Physical activity assessment (objective) T3 | 6 months follow-up
  Actigraph accelerometer at hip (Barnett et al., 2016): this is an objective measure of physical activity level, frequently used in physical activity studies with older adults. Participants will be asked to wear this accelerometer during seven days (day and night). They will be asked to register when and why they did not wear the device in a personal diary provided by the researchers.
Physical activity assessment (subjective) T4 | 12 months follow-up
  International Physical Activity Questionnaire - Short Form (IPAQ-SF) (Craig et al., 2003): this is an extensively used self-report measure for physical activity during the past seven days. It provides us with a categorical score of physical activity, distinguishing between low, moderate and high levels of physical activity.
Physical activity assessment (objective) T4 | 12 months follow-up
  Actigraph accelerometer at hip (Barnett et al., 2016): this is an objective measure of physical activity level, frequently used in physical activity studies with older adults. Participants will be asked to wear this accelerometer during seven days (day and night). They will be asked to register when and why they did not wear the device in a personal diary provided by the researchers.
General health questionnaires T1 - General Health | baseline
  The Patient-Reported Outcomes Measurement Information System (PROMIS) eight-item short form for General Health (Pellicciari et al., 2021): this is a self-report measure for global self-rated health with acceptable psychometric properties. This questionnaire provides us with a total score as well as distinct scores for mental and physical health.
  Scoring
  * PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  * A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured.
General health questionnaires T1 - Sleep Disturbances | baseline
  The Patient-Reported Outcomes Measurement Information System (PROMIS) four-item short form for Sleep Disturbances (Buysse et al., 2010; Terwee et al., 2014): this self-report measure with good psychometric properties assesses quality of sleep and prevalence of sleep difficulties.
  Scoring
  * PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  * A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured.
General health questionnaires T2 - General Health | 3 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) eight-item short form for General Health (Pellicciari et al., 2021): this is a self-report measure for global self-rated health with acceptable psychometric properties. This questionnaire provides us with a total score as well as distinct scores for mental and physical health.
  Scoring
  * PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  * A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured.
General health questionnaires T2 - Sleep Disturbances | 3 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) four-item short form for Sleep Disturbances (Buysse et al., 2010; Terwee et al., 2014): this self-report measure with good psychometric properties assesses quality of sleep and prevalence of sleep difficulties.
  Scoring
  * PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  * A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured.
General health questionnaires T3 - General Health | 6 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) eight-item short form for General Health (Pellicciari et al., 2021): this is a self-report measure for global self-rated health with acceptable psychometric properties. This questionnaire provides us with a total score as well as distinct scores for mental and physical health.
  Scoring
  * PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  * A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured.
General health questionnaires T3 - Sleep Disturbances | 6 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) four-item short form for Sleep Disturbances (Buysse et al., 2010; Terwee et al., 2014): this self-report measure with good psychometric properties assesses quality of sleep and prevalence of sleep difficulties.
  Scoring
  * PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  * A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured.
General health questionnaires T4 - General Health | 12 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) eight-item short form for General Health (Pellicciari et al., 2021): this is a self-report measure for global self-rated health with acceptable psychometric properties. This questionnaire provides us with a total score as well as distinct scores for mental and physical health.
  Scoring
  * PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  * A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured.
General health questionnaires T4 - Sleep Disturbances | 12 months follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) four-item short form for Sleep Disturbances (Buysse et al., 2010; Terwee et al., 2014): this self-report measure with good psychometric properties assesses quality of sleep and prevalence of sleep difficulties.
  Scoring
  * PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  * A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population.
  * For PROMIS measures, higher scores equals more of the concept being measured.

OTHER OUTCOMES:
Process evaluation questionnaire T1 | baseline,3 months, 6 months follow-up
  This will include questions on fidelity, delivered dose (completeness), received dose (exposure, satisfaction), participation rate, acceptability of the intervention, group dynamics, environmental context,…
Process evaluation questionnaire T2 | baseline,3 months, 6 months follow-up
  This will include questions on fidelity, delivered dose (completeness), received dose (exposure, satisfaction), participation rate, acceptability of the intervention, group dynamics, environmental context,…
Process evaluation questionnaire T3 | baseline,3 months, 6 months follow-up
  This will include questions on fidelity, delivered dose (completeness), received dose (exposure, satisfaction), participation rate, acceptability of the intervention, group dynamics, environmental context,…

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Hotterbeex, MSc, Principal Investigator — Ghent University / KU Leuven
Locations (2):
- Belgium (2):
  - Ghent University, Ghent, East-Flanders
  - KU Leuven, Leuven, Vlaams Brabant

IPD SHARING:
Plan to Share IPD: No